CLINICAL TRIAL: NCT01451996
Title: The Efficacy of Claritin in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16171A
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: direct-to-consumer advertising
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Claritin ads (Other): Subject will be given 10mg Claritin tablet and then watch a movie that includes commercials for Claritin.
  Interventions: Drug: Claritin
- Zyrtec ads (Other): Subject will be given 10mg Claritin tablet and then watch a movie that includes commercials for Zyrtec.
  Interventions: Drug: Claritin

INTERVENTIONS:
Drug: Claritin — Subject will be given 10mg Claritin tablet.

SUMMARY:
The primary goal of this study is to examine determinants of the efficacy of Claritin.

DETAILED DESCRIPTION:
Subjects will be given Claritin 10mg tablet. Subjects will be challenged with histamine via skin prick prior to Claritin administration and at 1 and 2 hours post administration. We will measure and record wheal and flare area 10 minutes following each challenge.

ELIGIBILITY:
Inclusion Criteria.

1. Males and females between 18 and 65 years of age.

Exclusion Criteria.

1. Pregnant or lactating women.
2. Upper respiratory infection within 14 days of study start.
3. Women of childbearing potential not using specific contraception method(s) (i.e., birth control pills, depo Provera, double barrier) as well as women who are breastfeeding.
4. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (heart, lung, kidney, neurological, oncologic or liver disease).
5. Use of any other investigational agent in the last 30 days.
6. Use of medications that may affect skin testing. Specifically, subjects are excluded if they have used an antihistamine during the 4 days preceding their treatment visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Malani, J.D., Ph.D, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Claritin Ads, Allergy+: Subject, with positive skin test to at least one common allergen (grass, trees, mold, dust mites, ragweed, cats), will be given 10mg Claritin tablet and then watch a movie that includes commercials for Claritin.
  Claritin: Subject will be given 10mg Claritin tablet.
- Zyrtec Ads, Allergy+: Subject, with positive skin test to at least one common allergen (grass, trees, mold, dust mites, ragweed, cats), will be given 10mg Claritin tablet and then watch a movie that includes commercials for Zyrtec.
  Claritin: Subject will be given 10mg Claritin tablet.
- Claritin Ads, Allergy-: Subject, without allergies, will be given 10mg Claritin tablet and then watch a movie that includes commercials for Claritin.
  Claritin: Subject will be given 10mg Claritin tablet.
- Zyrtec Ads, Allergy-: Subject, without allergies, will be given 10mg Claritin tablet and then watch a movie that includes commercials for Zyrtec.
  Claritin: Subject will be given 10mg Claritin tablet.
Period: Overall Study
Arm/Group | Claritin Ads, Allergy+ | Zyrtec Ads, Allergy+ | Claritin Ads, Allergy- | Zyrtec Ads, Allergy-
Started | 83 | 87 | 85 | 85
Completed | 83 | 87 | 85 | 85
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The sample was stratified into subjects with (Allergy+) and without (Allergy-) a positive skin test and block-randomized each subpopulation to the two advertisement conditions (Claritin ads and Zyrtec ads)
Groups:
- Total: Total of all reporting groups
Arm/Group | Claritin Ads, Allergy+ | Zyrtec Ads, Allergy+ | Claritin Ads, Allergy- | Zyrtec Ads, Allergy- | Total
Number analyzed (Participants) | 83 | 87 | 85 | 85 | 340
Age, Continuous [Mean (Full Range); unit: years] | 27.83 [18 to 65] | 29.30 [18 to 65] | 27.25 [18 to 65] | 26.40 [18 to 65] | 27.70 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 51 | 59 | 59 | 212
  Male | 40 | 36 | 26 | 26 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 29 | 35 | 24 | 22 | 110
  Not Black | 54 | 52 | 61 | 63 | 230
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 87 | 85 | 85 | 340

OUTCOME MEASURES:

1. Primary Outcome: Change in Wheal Reaction Area From Baseline --- 2 Hour
Description: A research technician, blinded to the subject's condition, measured the extent of the skin inflammation at baseline and 2 hours post Claritin administration by tracing the wheal reaction after the histamine challenge (i.e. the slightly reddened, elevated area at the site of the challenge, a well-established measure of histamine response). The percentage change in the wheal reaction was calculated as the change (decrease) in the size relative to baseline, multiplied by 100. Wheal area was measured in mm^2.
Time Frame: baseline and 2 hours post administration of Claritin.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Claritin Ads, Allergy+ | Zyrtec Ads, Allergy+ | Claritin Ads, Allergy- | Zyrtec Ads, Allergy-
Number analyzed (Participants) | 83 | 87 | 85 | 85
Percent change | 27.5 (2.5) | 29.0 (2.5) | 30.97 (2.4) | 25.0 (2.5)

2. Secondary Outcome: Change in Wheal Reaction Area From Baseline --- 1 Hour
Description: A research technician, blinded to the subject's condition, measured the extent of the skin inflammation at baseline and 1 hour post Claritin administration by tracing the wheal reaction after the histamine challenge (i.e. the slightly reddened, elevated area at the site of the challenge, a well-established measure of histamine response). The percentage change in the wheal reaction was calculated as the change (decrease) in the size relative to baseline, multiplied by 100. Wheal area was measured in mm^2.
Time Frame: baseline and 1 hours post administration of Claritin
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Claritin Ads, Allergy+ | Zyrtec Ads, Allergy+ | Claritin Ads, Allergy- | Zyrtec Ads, Allergy-
Number analyzed (Participants) | 83 | 87 | 85 | 85
Percent change | 10.8 (2) | 17.5 (2.5) | 14.18 (3) | 10.83 (3)

ADVERSE EVENTS:
Time Frame: 2 hours post Claritin use
Arm/Group | Claritin Ads, Allergy+ | Zyrtec Ads, Allergy+ | Claritin Ads, Allergy- | Zyrtec Ads, Allergy-
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/87 | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/83 | 0/87 | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes